CLINICAL TRIAL: NCT06617819
Title: Influence of Different Prostheses(CR Vs. PS) on Postoperative Clinical Functional Scores in Total Knee Arthroplasty Based on Extramedullary Femoral Osteotomy Techniques and Functionalist Alignment
Brief Title: Influence of Different Prostheses on Postoperative Clinical Function in Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Xu Zhihong, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-6668-01
Record Dates: First submitted 2024-09-22; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Knee Arthropathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- experimental group (Experimental): CR prosthesis for the left knee
  Interventions: Device: CR prosthesis
- control group (Active Comparator): PS prosthesis for the left knee
  Interventions: Device: PS prosthesis

INTERVENTIONS:
Device: CR prosthesis — For patients undergoing simultaneous bilateral knee arthroplasty, different prostheses (CR vs. PS) were randomized to the left or right knee.
  Arms: experimental group
Device: PS prosthesis — For patients undergoing simultaneous bilateral knee arthroplasty, different prostheses (CR vs. PS) were randomized to the left or right knee.
  Arms: control group

SUMMARY:
Exploring differences in knee function after surgery with different types of prostheses(Cruciate ligament retaining(CR) VS. posterior stabilizing(PS))

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-80 years, any gender, BMI < 35 kg/m2
2. Initial diagnosis of bilateral knee OA (Kellgren-Lawrence classification grades 3 or 4). Patients who are to undergo simultaneous primary bilateral knee arthroplasty
3. Inversion deformity ≤ 15°
4. Posterior cruciate ligament integrity

Exclusion Criteria:

1. History of knee surgery (ligament, osteotomy, etc.)
2. knee flexion<90°.
3. flexion contracture of one knee > 10°
4. Comorbidity with other diseases, such as peripheral neuropathy, malignant tumors, rheumatism, etc.
5. Posterior cruciate ligament injury
6. Those assessed to be intolerant of surgery

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee Society Score, KSS | 6 weeks, 3 months, 6 months, 12 months, 24 months after surgery
  Use of Knee Society Score scales for assessment. Including pain, mobility, stability, the patient's ability to walk, up and down the stairs, etc. on the assessment, 85-100 is excellent, 70-84 is good, 60-69 is pass, less than 60 is poor

SECONDARY OUTCOMES:
WOMAC | Preoperative, 6 weeks, 3 months, 6 months, 12 months, 24 months after surgery
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a composite outcome measure consisting of multiple measures: pain, stiffness and physical function. The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Stride length | Preoperative, 6 weeks, 3 months, 6 months, 12 months, 24 months after surgery
  The step length data were collected using a gait analysis instrument to analyze whether there was a difference between the right and left sides.
Stride frequency | Preoperative, 6 weeks, 3 months, 6 months, 12 months, 24 months after surgery
  The step frequency data were collected using an instrument to analyze whether there were any differences.
Percentage of stance phase | Preoperative, 6 weeks, 3 months, 6 months, 12 months, 24 months after surgery
  The stance phase is the time during which the lower limbs are in contact with the ground and are subjected to gravity, and accounts for 60% of the walking cycle. In walking disorders, the prolongation of the stance phase is often associated with impaired walking.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Xu, Doctor, Principal Investigator — Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University
Locations (1):
- Nanjing Drum Tower Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
IPD will be available by consulting the principal investigator